CLINICAL TRIAL: NCT03070639
Title: Enhancing Safe Sleep Practices of Urban Low-Income Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HD072821; 1R01HD072821-01A1 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Sudden Infant Death Syndrome
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Care Study Condition (No Intervention): The Standard of Care control group will not receive any additional services at the newborn visit.
- Attention-Matched Control Condition (Active Comparator): The Attention-Matched Control Condition will include the Scald Prevention Intervention.
  Interventions: Behavioral: Scald Prevention Intervention
- Safe Sleep Intervention Condition (Experimental): The Intervention Condition will include the Safe Sleep Intervention.
  Interventions: Behavioral: Safe Sleep Intervention

INTERVENTIONS:
Behavioral: Safe Sleep Intervention — A health educator will visit participant during their 2-week well visit in the clinic, to deliver a tailored intervention based on the baby's sleep practices. Participant will also receive a free pack'n play, sleep sack, and educational resources on safe sleep.
  Arms: Safe Sleep Intervention Condition
Behavioral: Scald Prevention Intervention — A health educator will visit participant during their 2-week well visit in the clinic, to deliver a tailored intervention based on practices regarding scald risks in the home. Participant will also receive a bath thermometer, candy/frying thermometer, and educational resources on scald prevention.
  Arms: Attention-Matched Control Condition

SUMMARY:
The specific aims of the study are to: 1) evaluate the impact of the safe sleep intervention on parents' knowledge, beliefs, intentions, skills and practices related to creating and maintaining a safe sleep environment for their infants during the first four months of life; 2) describe the characteristics of physician anticipatory guidance about safe sleep and identify physician, patient and parent characteristics associated with coverage of the topic at the well-child visits; and 3) evaluate the dissemination of the B'more for Healthy Babies (BHB)'s safe sleep campaign messages and services among our study participants.

DETAILED DESCRIPTION:
This intervention trial uses a randomized controlled design and will be conducted in the Harriet Lane Clinic. The study conditions are: Standard Care Group (SG), Attention-Matched Control Group that receives a scald burn prevention intervention (CG), and Intervention Group that receives a safe sleep intervention (IG). Parents or legal guardians will be enrolled during the newborn visit (when the baby is approximately 4-7 days old). While waiting to be seen for their 2-week well-child visit, the parent will complete the Baseline Interview and be randomized to SG, IG, or CG. All participants will receive Standard of Care during all of their well-child visits, which will include standard anticipatory guidance delivered by the pediatric resident. The IG and CG interventions will be delivered in the clinic during the 2-week visit after the baseline survey has been completed. The first follow-up will be conducted at the home of the parent after completing the 2-week visit, when the baby is approximately 3-6 weeks old. The second follow-up will be conducted at the home of the parent after the 2-month well-child visit, when the child is approximately 2-4 months of age. Each home visit consists of an interview covering safe sleep and scald topics, an observation of the baby's sleep environment, and testing the water temperature. The 2-week and 2-month well-child visits will be audio-recorded, and parent or legal guardians will be asked to complete a Visit Exit Checklist.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age) or emancipated minor.
* Parent or legal guardian of the child.
* Child is receiving care at the Harriet Lane Clinic.
* Child's primary care provider is participating in the study.
* English-speaking.
* Lives in Baltimore City or Baltimore County.
* Not homeless or not living in a shelter or in an established transitional housing facility.

Exclusion Criteria:

* Not an adult or emancipated minor.
* Not the parent or legal guardian of the child.
* Child is not receiving care at the Harriet Lane Clinic.
* Child's primary care provider is not participating in the study.
* Non English-speaker.
* Does not live in Baltimore City or Baltimore County.
* Homeless or living in a shelter or other established transitional housing facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the Effect of a Safe Sleep Intervention on the Safe Sleep Environment of Infants | Follow-up #1 (3-6 weeks)
  Assessed with a 125-item questionnaire.

SECONDARY OUTCOMES:
Evaluate the Effect of a Scald Prevention Intervention on Potential Scald Risks in the Home | Follow-up #1 (3-6 weeks)
  Assessed with a 45-item questionnaire.
Describe Characteristics of Physician Anticipatory Guidance on Safe Sleep and Other Safety Topics | 2-week well-child visit and 2-month well-child visit
  Assessed with an 11-item coding sheet and transcription file.

OTHER OUTCOMES:
Evaluate Dissemination of City Health Department's Safe Sleep Campaign Messages and Services Among Participants | Baseline survey (2 weeks)
  Assessed with a 13-item questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C Gielen, ScD, ScM, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Harriet Lane Clinic, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burrell TD, McDonald EM, Mahoney P, Musci RJ, Shields W, Gielen A, Solomon BS. Content of Infant Safe Sleep Counseling and Maternal Reported Practices in an Urban Clinic. Acad Pediatr. 2019 Sep-Oct;19(7):801-807. doi: 10.1016/j.acap.2019.06.014. Epub 2019 Jun 26. PMID 31254631
- [Derived] McDonald EM, Davani A, Price A, Mahoney P, Shields W, Musci RJ, Solomon BS, Stuart EA, Gielen AC. Health education intervention promoting infant safe sleep in paediatric primary care: randomised controlled trial. Inj Prev. 2019 Jun;25(3):146-151. doi: 10.1136/injuryprev-2017-042421. Epub 2017 Sep 22. PMID 28939661